CLINICAL TRIAL: NCT05649137
Title: Effect and Safety of Semaglutide 7.2 mg Once-weekly in Participants With Obesity and Type 2 Diabetes
Brief Title: A Research Study to See How Semaglutide Helps People With Excess Weight and Type 2 Diabetes Lose Weight
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9536-7545; 2022-002235-60 (EudraCT Number); U1111-1279-0359 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Obesity; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Semaglutide 7.2 mg (Experimental): Participants will receive once-weekly injection of semaglutide subcutaneously (s.c.) in 20 week dose escalation period with dose escalation (0.25 milligram [mg], 0.5 mg, 1.0 mg, 1.7 mg, 2.4 mg, and 7.2 mg) every fourth week. Treatment will be continued on the maintenance dose of 7.2 mg once-weekly for an additional 52 weeks until week 72.
  Interventions: Drug: Semaglutide
- Semaglutide 2.4 mg (Experimental): Participants will receive once-weekly s.c. injection of semaglutide in 20 week dose escalation period with dose escalation (0.25 mg, 0.5 mg, 1.0 mg, 1.7 mg, and 2.4 mg) every fourth week until maintenance dose of 2.4 mg of semaglutide was reached. Treatment will be continued on the maintenance dose of 2.4 mg once-weekly for an additional 52 weeks until week 72.
  Interventions: Drug: Semaglutide
- Placebo (Placebo Comparator): Participants will receive once-weekly s.c. injection of placebo matched to semaglutide for 72 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide — Participants will receive once-weekly s.c. injections of semaglutide in escalating doses (0.25 mg, 0.5 mg, 1.0 mg, 1.7 mg, 2.4 mg and 7.2 mg) every fourth week. Treatment will be continued on the maintenance dose of 7.2 mg once-weekly for an additional 52 weeks. Injections may be administered in the thigh, abdomen, or upper arm, at any time of day irrespective of meals.
  Arms: Semaglutide 7.2 mg
Drug: Semaglutide — Participants will receive once-weekly s.c. injections of semaglutide in escalating doses (0.25 mg, 0.5 mg, 1.0 mg, 1.7 mg, and 2.4 mg) every fourth week. Treatment will be continued on the maintenance dose of 2.4 mg once-weekly for an additional 52 weeks. Injections may be administered in the thigh, abdomen, or upper arm, at any time of day irrespective of meals.
  Arms: Semaglutide 2.4 mg
Drug: Placebo — Participants will receive once-weekly s.c. injection of placebo matched to semaglutide for 72 weeks. Injections may be administered in the thigh, abdomen, or upper arm, at any time of day irrespective of meals.
  Arms: Placebo

SUMMARY:
This study will look at how much weight participants will lose and how much blood sugar control they achieve from the start to the end of the study. The weight loss in participants taking the investigational high dose of semaglutide will be compared to the weight loss in people taking "dummy" medicine and a lower dose of semaglutide. In addition to taking the medicine, participants will have talks with study staff about healthy food choices and how to be more physically active. Participants will either get semaglutide or "dummy" medicine. Which treatment participants get is decided by chance. Participants are more likely (4 out of 5) to get semaglutide than the "dummy" medicine. The study medicine will be injected briefly, under skin, with a thin needle, typically in the stomach, thighs, or upper arms. After receiving first dose, the dose of semaglutide will be gradually increased until reaching the target dose. The study will last for about 1.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Age above or equal to 18 years at the time of signing informed consent.
* BMI greater than or equal to 30.0 kilograms per square meter (kg/m^2).
* Diagnosed with type 2 diabetes (T2D) greater than or equal to 180 days prior to the day of screening.
* History of at least one self-reported unsuccessful dietary effort to lose body weight.
* HbA1c 7.0-10.0 percent (53-86 millimoles per mole [mmol/mol]) (both inclusive) as measured by central laboratory at screening.

Exclusion Criteria:

* A self-reported change in body weight greater than 5 kilograms (kg) (11 pounds [lbs]) within 90 days before screening irrespective of medical records.
* Personal or first-degree relative(s) history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma.
* Renal impairment with estimated Glomerular Filtration Rate (eGFR) less than 30 milliliters per minute per 1.73 square meter (30 mL/min/1.73 m^2) (less than 45 mL/min/1.73 m^2 in participants treated with Sodium-glucose Cotransporter-2 [SGLT2i]) according to Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine equation as defined by Kidney Disease: Improving Global Outcomes (KDIGO) 2012 by the central laboratory at screening.
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within 90 days before screening or in the period between screening and randomization. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2023-01-04 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Semaglutide 7.2 mg versus Placebo: Relative change in body weight | From baseline (week 0) to end of treatment (week 72)
  Measured in percentage (%).
Semaglutide 7.2 mg versus Placebo: Number of participants who achieve body weight reduction greater than or equal to (>=) 5% (yes/no) | From baseline (week 0) to end of treatment (week 72)
  Measured as count of participants.

SECONDARY OUTCOMES:
Semaglutide 7.2 mg versus Placebo: Number of participants who achieve body weight reduction >=10% (yes/no) | From baseline (week 0) to end of treatment (week 72)
  Measured as count of participants.
Semaglutide 7.2 mg versus Placebo: Number of participants who achieve body weight reduction >=15% (yes/no) | From baseline (week 0) to end of treatment (week 72)
  Measured as count of participants.
Semaglutide 7.2 mg versus Placebo: Number of participants who achieve body weight reduction >=20% (yes/no) | From baseline (week 0) to end of treatment (week 72)
  Measured as count of participants.
Semaglutide 7.2 mg versus Placebo: Change in waist circumference | From baseline (week 0) to end of treatment (week 72)
  Measured in centimeters (cm).
Semaglutide 7.2 mg versus Placebo: Change in glycated haemoglobin (HbA1c) | From baseline (week 0) to end of treatment (week 72)
  Measured in percentage (%).
Semaglutide 7.2 mg versus Placebo: Change in body weight | From baseline (week 0) to end of treatment (week 72)
  Measured in kilograms (kg).
Semaglutide 7.2 mg versus Placebo: Change in body mass index (BMI) | From baseline (week 0) to end of treatment (week 72)
  Measured in kilograms per square meter (kg/m^2).
Semaglutide 7.2 mg versus Placebo: Change in systolic blood pressure | From baseline (week 0) to end of treatment (week 72)
  Measured in millimeters of mercury (mmHg).
Semaglutide 7.2 mg versus Placebo: Change in diastolic blood pressure | From baseline (week 0) to end of treatment (week 72)
  Measured in mmHg.
Semaglutide 7.2 mg versus Placebo: Change in total cholesterol | From baseline (week 0) to end of treatment (week 72)
  Measured in ratio to baseline.
Semaglutide 7.2 mg versus Placebo: Change in high-density lipoprotein (HDL) cholesterol | From baseline (week 0) to end of treatment (week 72)
  Measured in ratio to baseline.
Semaglutide 7.2 mg versus Placebo: Change in low-density lipoprotein (LDL) cholesterol | From baseline (week 0) to end of treatment (week 72)
  Measured in ratio to baseline.
Semaglutide 7.2 mg versus Placebo: Change in very-low-density lipoprotein (VLDL) cholesterol | From baseline (week 0) to end of treatment (week 72)
  Measured in ratio to baseline.
Semaglutide 7.2 mg versus Placebo: Change in triglycerides | From baseline (week 0) to end of treatment (week 72)
  Measured in ratio to baseline.
Semaglutide 7.2 mg versus Placebo: Change in free fatty acids | From baseline (week 0) to end of treatment (week 72)
  Measured in ratio to baseline.
Semaglutide 7.2 mg versus Placebo: Change in high-sensitivity c reactive protein (hsCRP) | From baseline (week 0) to end of treatment (week 72)
  Measured in ratio to baseline.
Semaglutide 7.2 mg versus Placebo: Change in fasting plasma glucose | From baseline (week 0) to end of treatment (week 72)
  Measured in milligrams per deciliter (mg/dL).
Semaglutide 7.2 mg versus Placebo: Change in fasting serum insulin | From baseline (week 0) to end of treatment (week 72)
  Measured in ratio to baseline.
Semaglutide 7.2 mg versus Placebo: Number of participants with HbA1c less than (<) 7.0% (53 millimoles per mole [mmol/mol]) | From baseline (week 0) to end of treatment (week 72)
  Measured as count of participants.
Semaglutide 7.2 mg versus Placebo: Number of participants with HbA1c less than or equal to (<=) 6.5 % (48 mmol/mol) | From baseline (week 0) to end of treatment (week 72)
  Measured as count of participants.
Semaglutide 7.2 mg versus Placebo: Number of adverse events (AEs) | From baseline (week 0) to end of study (week 81)
  Measured as count of events.
Semaglutide 7.2 mg versus Placebo: Number of serious adverse events (SAEs) | From baseline (week 0) to end of study (week 81)
  Measured as count of events.
Semaglutide 7.2 mg versus Placebo: Change in pulse | From baseline (week 0) to end of treatment (week 72)
  Measured in beats per minute (bpm).
Semaglutide 7.2 mg versus Placebo: Number of treatment emergent severe or blood glucose confirmed symptomatic hypoglycaemic episodes | From baseline (week 0) to end of study (week 81)
  Measured as count of episodes.
Semaglutide 7.2 mg versus Semaglutide 2.4 mg: Number of AEs | From baseline (week 0) to end of study (week 81)
  Measured as count of events.
Semaglutide 7.2 mg versus Semaglutide 2.4 mg: Number of SAEs | From baseline (week 0) to end of study (week 81)
  Measured as count of events.
Semaglutide 7.2 mg versus Semaglutide 2.4 mg: Number of treatment emergent severe or blood glucose confirmed symptomatic hypoglycaemic episodes | From baseline (week 0) to end of study (week 81)
  Measured as count of episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (68):
- United States (21):
  - Univ of Alabama Birmingham, Birmingham, Alabama
  - John Muir Physicians Network, Concord, California
  - Velocity Clinical Research Westlake, Los Angeles, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - New West Physicians PC, Golden, Colorado
  - ARS- Deland CRU, DeLand, Florida
  - Jacksonville Ctr for Clin Res, Jacksonville, Florida
  - Florida Inst For Clin Res LLC, Orlando, Florida
  - Oviedo Medical Research, LLC, Oviedo, Florida
  - Hope Clin Res & Wellness, Conyers, Georgia
  - University of North Carolina, Chapel Hill, North Carolina
  - PharmQuest Life Sciences LLC, Greensboro, North Carolina
  - Amarillo Med Spec LLP, Amarillo, Texas
  - Elligo Clin Res Centre, Austin, Texas
  - Velocity Clin Res, Dallas, Dallas, Texas
  - UT Southwestern Medical Center - Lingvay, Dallas, Texas
  - PlanIt Research, PLLC, Houston, Texas
  - DCOL Ctr for Clin Res, Longview, Texas
  - Sugar Lakes Family Practice PA, Sugar Land, Texas
  - National Clin Res Inc., Richmond, Virginia
  - Selma Medical Associates, Winchester, Virginia
- Bulgaria (9):
  - "MHAT-Blagoevgrad", Department of Internal Diseases, Blagoevgrad
  - IPSOMC - Dr. Georgi Marinov, Burgas
  - "Medical Center Viva Feniks" Ood, Dobrich
  - UMHAT Pulmed, Department of endocrinology, Pazardzhik
  - 'MHAT Sveta Karidad' EAD, Plovdiv
  - 'MHAT Hadzhi Dimitar' OOD, Sliven
  - DCC VII - Sofia EOOD, Endocrinology, Sofia
  - "UMHAT- Prof. dr. Stoyan Kirkovich", Stara Zagora
  - "MHAT "Sveti Panteleimon" - Yambol" AD, Yambol
- Canada (6):
  - Ocean West Research Clinic, Surrey, British Columbia
  - G.A. Research Associates Ltd., Moncton, New Brunswick
  - Nova Scotia Hlth Halifax, Halifax, Nova Scotia
  - Premier Clinical Trial Research Network (PCTRN), Hamilton, Ontario
  - Wharton Med Clin Trials, Hamilton, Ontario
  - Milestone Research, London, Ontario
- Hungary (7):
  - Lausmed Kft., Baja, Bács-Kiskun county
  - Belinus Bt., Debrecen, Hajdú-Bihar
  - Borbánya Praxis E.Ü. Kft., Nyíregyháza, Szabolcs-Szatmar Varmegye
  - ClinDiab Egészségügyi Szolgáltató és Kereskedelmi Kft., Budapest
  - Bajcsy-Zsilinszky Kórház, Budapest
  - MED-TIMA Kft., Budapest
  - Fejér Megyei Szent György Oktatókórház, Székesfehérvár
- Poland (7):
  - Med. Cent. Diabet. Endo. Metabol. DIAB-ENDO-MET, Krakow, Lesser Poland Voivodeship
  - NZOZ Przychodnia Specjalistyczna Medica, Lublin, Lubelski
  - NZOZ "CenterMed Lublin" Sp. z o.o., Lublin, Lublin Voivodeship
  - Kresmed Sp. z o. o., Bialystok, Podlaskie Voivodeship
  - Uniwersyteckie Centrum Kliniczne SUM w Katowicach, Katowice
  - NBR Polska Tomasz Klodawski, Warsaw
  - PANSTWOWY INSTYTUT MEDYCZNY MSWiA, Warsaw
- Portugal (3):
  - Unidade Local De Saude De Matosinhos E.P.E., Senhora Da Hora, Matosinhos, Matosinhos
  - APDP - Associação Protectora dos Diabéticos de Portugal, Lisbon
  - Unidade Local de Saude de Sao Joao E.P.E, Porto
- Slovakia (6):
  - DIADA s.r.o., Bardejov
  - DIADA, s.r.o., Bardejov
  - Diab - Int, s.r.o., Bytča
  - ENDOMED, s.r.o., Košice
  - MED-DIA CENTRUM s.r.o., Považská Bystrica
  - DIABETOL, s.r.o., Prešov
- South Africa (9):
  - Phoenix Pharma, Port Elizabeth, Eastern Cape
  - Medi-Clinic Bloemfontein, Bloemfontein, Free State
  - Deepak Lakha, Johannesburg, Gauteng
  - Hemant Makan, Johannesburg, Gauteng
  - Wits Bara Clinical Trial Site, Johannesburg, Gauteng
  - Maxwell Centre, Durban, KwaZulu-Natal
  - Dr N.K. Gounden Medical Centre, Durban, KwaZulu-Natal
  - Lenmed Shifa Private Hospital, Durban, KwaZulu-Natal
  - Dr T Padayachee, eMkhomazi, KwaZulu-Natal

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisktrials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Lingvay I, Bergenheim SJ, Buse JB, Freitas P, Garvey WT, Harder-Lauridsen NM, Rosenstock J, Sahu K, Wharton S; STEP UP T2D trial group. Once-weekly semaglutide 7.2 mg in adults with obesity and type 2 diabetes (STEP UP T2D): a randomised, controlled, phase 3b trial. Lancet Diabetes Endocrinol. 2025 Nov;13(11):935-948. doi: 10.1016/S2213-8587(25)00225-6. Epub 2025 Sep 14. PMID 40961953